CLINICAL TRIAL: NCT03169335
Title: A Multi-center, Randomized, Double-blind, Parallel, Two-group Phase III Clinical Study of the Efficacy and Safety of QL1101 and Avastin® Respectively Combined With Paclitaxel and Carboplatin in the First-line Treatment of Non-squamous Non-small Cell Lung Cancer
Brief Title: Efficacy and Safety of QL1101 and Avastin® Respectively Combined With Paclitaxel and Carboplatin in the First-line Treatment of Non-squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QL1101-002
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2017-05

CONDITIONS: Non-squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Bevacizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): QL1101 + paclitaxel/carboplatin:subjects are given 15 mg/kg QL1101 on Day 1 of each cycle with every 3 weeks as a cycle, respectively combined with paclitaxel/carboplatin for 6 cycles (at least 4 cycles).
  Interventions: Drug: QL1101; Drug: Paclitaxel; Drug: Carboplatin
- Control group (Active Comparator): Avastin® + paclitaxel/carboplatin:subjects are given 15 mg/kg Avastin® on Day 1 of each cycle with every 3 weeks as a cycle, respectively combined with paclitaxel/carboplatin for 6 cycles (at least 4 cycles).
  Interventions: Drug: Avastin®; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: QL1101 — targeted vascular endothelial growth factor (VEGF) monoclonal antibodies
  Arms: Experimental group
Drug: Avastin® — targeted vascular endothelial growth factor (VEGF) monoclonal antibodies
  Other Names: bevacizumab
  Arms: Control group
Drug: Paclitaxel — 175 mg/m2, IV (in the vein) following investigational product on day 1 of each 21 day cycle. Number of cycles 4-6.
Drug: Carboplatin — AUC 5 IV, (in the vein) following paclitaxel on day 1 of each 21 day cycle. Number of cycles: 4-6.

SUMMARY:
The objective of this study is to assess the similarity between QL1101 and Avastin® respectively combined with chemotherapy in terms of efficacy and safety in patients with non-squamous non-small cell lung cancer. The study intends to include first-line patients with non-squamous non-small cell lung cancer, and uses QL1101 combined with basic chemotherapy CP (paclitaxel + carboplatin). The regimen is consistent with the usage and dosage of Avastin® at home and abroad indicated for the treatment of non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, positive drug-controlled, multi-center Phase III study. It is planned to enroll 512 treatment-naïve patients with non-squamous non-small cell lung cancer (NSCLC). Subjects are randomized into the QL1101 combined with paclitaxel/carboplatin or Avastin® combined with paclitaxel/carboplatin treatment group by a ratio of 1:1, and stratified by age (≥65 years, <65 years), sex (male, female) and EGFR subtype (sensitive mutation type, wild type).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and ≤75 years; 2) Patients with histologically or cytologically confirmed inoperable locally advanced (Stage IIIb, not suitable for multidisciplinary treatment), metastatic (Stage IV), or relapsed non-squamous cell non-small cell lung cancer. Diagnostic result of non-squamous cell non-small cell lung cancer obtained based on sputum cytology should be immunohistochemically confirmed. If a variety of tumor ingredients are mixed, the main cell types should be classified;
* ECOG score of 0-1 points;
* At least one measurable lesion can be evaluated according to RECIST1.1 criteria; Lesions situated in a previously irradiated area are considered measurable only if marked progressive signs occur after irradiation
* Patients who have not received systemic anti-tumor therapy of locally advanced or metastatic non-squamous non-small cell lung cancer (if the subject received adjuvant therapy after completing the radical treatment of early non-small cell lung cancer, but then the disease relapsed, the subject can be enrolled. In this case, the end time of the adjuvant therapy is required to be more than 6 months from the time of the first administration of this study, and various toxic reactions resulting from the adjuvant therapy should have recovered (≤ Grade 1 by CTCAE 4.03 criteria, except for alopecia).
* Expected survival time ≥24 weeks.
* Subjects must give informed consent to this study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

* Central squamous cell carcinoma, and mixed gland squamous cell carcinoma with squamous cell as the main ingredient;
* ALK fusion gene is known to be positive;
* Medical history or examination shows thrombotic disease within 6 months prior to screening;
* Imaging shows signs of tumor invasion of large vessels, and the investigator or radiologist must exclude patients whose tumor has been completely close to or surrounded or invaded the lumen of large vessels (e.g., the superior pulmonary artery or superior vena cava);
* Patients with a past history of symptomatic brain metastases or meningeal metastases, or spinal cord compression;
* Patients who received palliative radiotherapy for bone lesions outside the chest within 2 weeks prior to the first dose of the study drug;
* Patients who received major surgical procedures (including thoracotomy), or suffered from major trauma (such as fractures) within 28 days prior to screening, or need to undergo major surgery during the expected study treatment period;
* Patients who received a minor surgical procedure within 48 hours prior to the first treatment with Anivitis®/QL1101 (the investigator judges whether there is bleeding tendency);
* Patients who are currently using or have recently used (within 10 days prior to the first dose of Avastin®/QL1101) aspirin (>325 mg/day) or other nonsteroidal antiinflammatory drugs known to inhibit platelet function, or full-dose anticoagulants;
* Patients whose medical history or examination shows hereditary bleeding tendency or coagulation disorders, which may increase the risk of bleeding; -Uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg);
* Patients who had a past history of hypertensive crisis or hypertensive encephalopathy;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 18 weeks
  The actual endpoint is best response seen during the study

SECONDARY OUTCOMES:
Disease control rate | 3 months, 6 months, 9 months, 1 year
  DOR is defined as the time from the first tumor evaluation as CR or PR to the first evaluation as PD or death
Overall survival (OS) | 18 months after enrollment and randomization of the last case
  OS is defined as the time from randomization and grouping to patient death due to various causes. For patients who are lost to follow-up, the date when they were contacted for the last time will be used as the cut off time.
Progression-free survival (PFS) | 18 months after enrollment and randomization of the last case
  PFS is defined as the time from randomization and grouping to PD or death.
Treatment-emergent adverse events | 18 weeks
  Assessment following therapy with either QL1101 or avastin

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Chest hospital, Shanghai
  - Tianjin Chest hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Undecided